CLINICAL TRIAL: NCT06140134
Title: A Single-Arm Nonrandomized Phase II Study of Liver Transplantation in Locally Advanced Unresectable Non-Metastatic Intrahepatic Cholangiocarcinoma Treated With Neoadjuvant Systemic Therapy
Brief Title: Liver Transplantation in Intrahepatic Cholangiocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Keri E. Lunsford, Director of Translational and Surgical Science, Department of Surgery/Assistant Professor, Division of Transplant and Hepatobiliary Surgery/Member, Center for Immunity and Inflammation, Rutgers, The State University of New Jersey
Other Study IDs: Pro2021000973
Record Dates: First submitted 2023-10-02; First posted 2023-11-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Intrahepatic Cholangiocarcinoma; Cholangiocarcinoma, Intrahepatic
Keywords: liver transplantation; neoadjuvant systemic therapy; intrahepatic cholangiocarcinoma; iCCA; locally advanced non-metastatic iCCA; non-metastatic intrahepatic cholangiocarcinoma; liver transplant; unresectable intrahepatic cholangiocarcinoma; locally advanced intrahepatic cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Serial collection of patient blood for fractionation into serum/plasma and PBMCs (peripheral blood mononuclear cells) will be cryopreserved. Liver explant tissue (tumor and non-tumor) and biopsy samples will be collected. Samples will be utilized for extraction of DNA, RNA, protein, and histologic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intrahepatic cholangiocarcinoma listed for liver transplant: Listed patients enrolled with diagnosis of intrahepatic cholangiocarcinoma will be enrolled on an intent to treat basis with comparison between patients receiving transplant versus those who expire or are removed from the waitlist.
  Interventions: Procedure: Liver Transplant

INTERVENTIONS:
Procedure: Liver Transplant — Whole liver allotransplantation will be performed for patients on the liver transplant waiting list
  Other Names: Orthotopic liver transplantation

SUMMARY:
The aim of the current study is to determine the potential efficacy of liver transplantation in the form of patients' overall survival (OS) after neoadjuvant systemic therapy in patients with biologically responsive locally advanced non-metastatic intrahepatic cholangiocarcinoma (iCCA) in comparison to patients historically treated with chemotherapy alone.

DETAILED DESCRIPTION:
Research Significance:

Cholangiocarcinoma, which arises from biliary epithelium, can be anatomically subdivided into distal, hilar, and intrahepatic subgroups. Intrahepatic cholangiocarcinoma (iCCA) constitutes the second most common primary liver cancer after hepatocellular carcinoma, with a rising incidence but without parallel advances in treatment or patient outcome. At present, surgical resection is the only widely accepted potentially curative therapy for iCCA; however, 5-year survival rates for resectable disease are less than 25%. This high mortality is attributed to high tumor recurrence. Two-thirds of patients who undergo curative-intent resection for iCCA suffer from postoperative disease recurrence, most commonly in the remnant liver, followed by the peritoneum and abdominal lymph nodes. Approximately 83% of recurrences occur within the first 2 years after resection, suggesting inadequate local tumor control with resection in this highly infiltrative cancer.

Liver transplantation for intrahepatic cholangiocarcinoma:

While liver transplantation has been previously investigated for unresectable iCCA, the outcomes have been poor in comparison to the results for hepatocellular carcinoma, with 18-25% OS and RFS after 5 years; however, most studies evaluated patients with either incidental iCCA or iCCA misdiagnosed prior to transplant as hepatocellular carcinoma (HCC). Thus, iCCA is considered by most centers to be a formal contraindication to liver transplantation.

Neoadjuvant therapy with subsequent liver transplantation for perihilar cholangiocarcinoma:

Similar to iCCA, liver transplantation outcomes for perihilar cholangiocarcinoma were initially poor; however, an analysis of the United Network of Organ Sharing (UNOS) database found a significant survival benefit for patients with perihilar cholangiocarcinoma who received pre-transplant neoadjuvant systemic therapy compared with patients who transplanted for incident disease. Subsequently, several studies reported improved survival for hilar cholangiocarcinoma treated with neoadjuvant chemoradiation followed by liver transplantation. A multicenter study reported a 65% 5-year survival rate; liver transplantation has thus become the preferred treatment for patients with locally advanced unresectable hilar cholangiocarcinoma. Response to neoadjuvant therapy probably offers a means to select patients with hilar cholangiocarcinoma who might benefit from transplantation.

Neoadjuvant therapy with subsequent liver transplantation for intrahepatic cholangiocarcinoma (iCCA):

The published literature regarding liver transplantation (LT) for iCCA is mostly limited to incidental or misdiagnosed tumors identified on pathology, with most patients not receiving neoadjuvant therapy. Retrospective analysis including a small cohort of patients receiving neoadjuvant therapy showed that pre-transplant therapy appeared to decrease disease recurrence; however, reports did not distinguish between hilar cholangiocarcinoma and iCCA. In 2016, a multi-center, international, retrospective study investigated outcomes of liver transplantation in 48 iCCA patients who had not received neoadjuvant chemotherapy or locoregional therapy. In that study, 5-year OS was 65% for iCCA ≤2 cm and 45% for advanced larger lesions. Survival outcomes for locally advanced iCCA were worse, but patients having received pre-transplant neoadjuvant therapy in this series were excluded. The effect of neoadjuvant chemotherapy in patients with larger and multifocal tumors remains largely undefined. In 2020, another multicenter study compared the outcomes of patients with cirrhosis undergoing liver transplantation or liver resection who had iCCA or combined hepatocellular-cholangiocarcinoma (cHCC-CCA). The retrospective study analyzed a total of 49 LT and 26 liver resected patients with cirrhosis and histologically confirmed iCCA/ cHCC-CCA ≤5 cm. Results suggested that liver transplanted patients had a significantly lower tumor recurrence (diameter of largest nodule and tumor differentiation were independently predictive) and had a significantly higher 5-year recurrence-free survival. The effects of liver transplantation may provide a benefit for highly selected patients with cirrhosis and unresectable iCCA/cHCC-CCA with specific tumor dimensions. These findings suggests that liver transplantation might be a viable option for small, solitary iCCA in the absence of pre-transplant therapy or with locoregional therapy alone.

A subset of patients with iCCA experienced sustained response to neoadjuvant therapy, and it has been postulated that response duration might be an appropriate surrogate marker for the selection of patients for liver transplantation. Through the Methodist-MD Anderson Joint Cholangiocarcinoma Collaborative Committee, a recent prospective case-series of 6 patients with locally advanced unresectable iCCA without extrahepatic disease or vascular involvement was performed. Patients treated with neoadjuvant systemic chemotherapy with a minimum of 6 months radiographic disease stability or regression received liver transplantation. The median post-transplant follow-up duration was 36 months (range; 29-51). The OS rate was 100% (95% Confidence interval [CI]; 100-100) at 1-year, 83·3% (95% CI; 27·3-97·5) at 3 years, and 83·3% (95% CI; 27·3-97·5) at 5 years. Three patients developed post-transplant recurrence at a median of 7·6 months with 50% (95% CI; 11·1-80·4) RFS at 1-, 3-, and 5-years. Since publication, an additional 5 patients have been transplanted, and all patients have been followed for an additional 24 months. More recent data indicates a 5-year OS of 79.5% with RFS of 42.4%. In regards to recurrence, 4 of 5 occurred within 12 months of transplant. Retrospective evaluation of the pre-transplant imaging demonstrated evidence of pre-transplant extrahepatic disease. More stringent patient selection, such as the addition of a PET-CT scan, would likely avoid early recurrence in the majority of patients. Adverse events have been reported, including grade 3 postoperative ileus in one patient and grade 4 acute kidney injury requiring temporary dialysis in another patient. Both adverse events were among those commonly occurring with liver transplantation for any indication. No post-operative complications could be directly related to this protocol. Therefore, the investigators anticipate that selected patients with locally advanced non-metastatic iCCA who show pre-transplant disease stability on neoadjuvant therapy might benefit from liver transplantation.

Research Design and Methods:

This is a single-center phase II study. Patients with locally advanced unresectable iCCA with no evidence of vascular invasion or extrahepatic disease who have at least 6 months of disease stability or regression on neoadjuvant systemic therapy will be enrolled. Eligible patients who also meet center-specific medical criteria for transplant listing will be listed in the United Network of Organ Sharing (UNOS) national registry. When a decision is made to list the patient, the patient will be assigned a subject identification number. All organ offers will be received as per UNOS regulations. When a matching donor liver becomes available, the inclusion and exclusion criteria will be re-verified.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age on the day of consenting to the study.
* Patients must have histologically confirmed diagnosis of locally advanced intrahepatic cholangiocarcinoma
* Confirmed diagnosis of locally advanced unresectable iCCA with no vascular invasion, lymph node, or extrahepatic disease.
* Unresectable disease based on tumor location or underlying liver disease
* Patients must have ≥ 6 months of disease stability or tumor regression on neoadjuvant therapy. In cases in which patients had received second-line therapy, disease must also have been controlled for ≥ 6 months on that regimen.
* Patients who had previous surgical resection for iCCA are eligible if surgery occurred more than 6 months prior to listing, and patients have had ≥ 6 months of disease stability or response on therapy.
* ECOG performance status ≤1 (Karnofsky ≥70%, see Appendix A).
* Patients must have organ and marrow function acceptable for liver transplantation per institutional protocol:
* If history of chronic hepatitis B virus (HBV) infection, viral load should be undetectable on suppressive therapy.
* If history of chronic hepatitis C virus (HCV) infection, patients should have undetectable HCV viral load.
* Women of child-bearing years must have contraception plan in place from the time of study enrollment until at least one year following liver transplant.
* Ability to understand and the willingness to sign a written informed consent document
* Meets all other medical and psychosocial criteria for liver transplant
* Demonstrate ability to comply with study procedures

Exclusion Criteria:

* Age <18 years of age on the day of consenting to the study.
* Patients who have extrahepatic metastases, lymph node involvement, invasion or encasement of major hepatic vascular structures, perforation of the visceral peritoneum, invasion of extrahepatic structures, invasion of perihilar fat, periductular invasion, concurrent hepatoma or mixed hepatocellular cholangiocarcinoma.
* Concurrent severe and/or uncontrolled concurrent illness including, but not limited to, ongoing or active infection, acute fulminant liver failure, symptomatic congestive heart failure, unstable angina pectoris, severe uncorrected coronary artery disease, severe cerebrovascular disease, severe pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements and that would exclude the patient from eligibility for liver transplantation per institutional protocol.
* Prior solid organ or bone marrow transplant
* Dependent on ≥2 IV inotropic support to maintain hemodynamics
* Previous (within the past 5 years) or concurrent presence of other cancer, except non-melanoma skin cancer and in situ carcinomas.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Scale score >1 (Karnofsky <70%, see Appendix A).
* Unable to understand and sign a written informed consent document
* Untreated viral hepatitis
* Pregnant or breast-feeding women
* HIV-infected patients

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biologically responsive locally advanced non-metastatic intrahepatic cholangiocarcinoma (iCCA) treated with neoadjuvant systemic chemotherapy with a radiographic disease stability or regression.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
5-year Overall Survival Rate (ORS) | 5 years from the time of transplant or until death of patient, whichever came first
  5-year ORS is the length of time that patients diagnosed with locally advanced non-metastatic intrahepatic cholangiocarcinoma (iCCA) treated with neoadjuvant systemic therapy followed by liver transplant (LT) are still alive post-LT.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | From date of transplant until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  RFS is the length of time from liver transplantation (LT) to the time of disease recurrence, time of patient death, or time of study completion for patients with locally advanced non-metastatic intrahepatic cholangiocarcinoma treated with neoadjuvant systemic therapy followed by liver transplantation.
Intent-to-treat Overall Survival Rate (ITT ORS) | 5 years from time of waitlist or until death of patient, whichever came first
  ITT ORS is the length of time that patients diagnosed with locally advanced non-metastatic intrahepatic cholangiocarcinoma (iCCA) treated with neoadjuvant systemic therapy and waitlisted for liver transplant for iCCA are still alive after being waitlisted for liver transplantation.
Post-liver transplant functional assessments to identify postoperative complications, short-term morbidities, and long-term morbidities | From date of emergence of a post-transplant adverse event until the date the adverse event is designated as resolved by investigator or its effect on patient's condition stabilizes, whichever came first, assessed up to 5 years
  All serious adverse events will be followed and documented, including bleeding requiring re-operation, hepatic artery or portal vein thrombosis, bile duct leak, bile duct stricture, primary non-function of the transplant liver, need for re-transplant of the liver.

CONTACTS AND LOCATIONS:
Overall Officials: Keri E Lunsford, MD, PhD, Principal Investigator — Rutgers University
Locations (2):
- United States (2):
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - University Hospital, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study after deidentification (text, tables, figures and appendices)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Following publication of study results

REFERENCES:
- [Background] Banales JM, Cardinale V, Carpino G, Marzioni M, Andersen JB, Invernizzi P, Lind GE, Folseraas T, Forbes SJ, Fouassier L, Geier A, Calvisi DF, Mertens JC, Trauner M, Benedetti A, Maroni L, Vaquero J, Macias RI, Raggi C, Perugorria MJ, Gaudio E, Boberg KM, Marin JJ, Alvaro D. Expert consensus document: Cholangiocarcinoma: current knowledge and future perspectives consensus statement from the European Network for the Study of Cholangiocarcinoma (ENS-CCA). Nat Rev Gastroenterol Hepatol. 2016 May;13(5):261-80. doi: 10.1038/nrgastro.2016.51. Epub 2016 Apr 20. PMID 27095655
- [Background] Spolverato G, Kim Y, Ejaz A, Alexandrescu S, Marques H, Aldrighetti L, Gamblin TC, Pulitano C, Bauer TW, Shen F, Sandroussi C, Poultsides G, Maithel SK, Pawlik TM. Conditional Probability of Long-term Survival After Liver Resection for Intrahepatic Cholangiocarcinoma: A Multi-institutional Analysis of 535 Patients. JAMA Surg. 2015 Jun;150(6):538-45. doi: 10.1001/jamasurg.2015.0219. PMID 25831462
- [Background] Benson AB 3rd, Abrams TA, Ben-Josef E, Bloomston PM, Botha JF, Clary BM, Covey A, Curley SA, D'Angelica MI, Davila R, Ensminger WD, Gibbs JF, Laheru D, Malafa MP, Marrero J, Meranze SG, Mulvihill SJ, Park JO, Posey JA, Sachdev J, Salem R, Sigurdson ER, Sofocleous C, Vauthey JN, Venook AP, Goff LW, Yen Y, Zhu AX. NCCN clinical practice guidelines in oncology: hepatobiliary cancers. J Natl Compr Canc Netw. 2009 Apr;7(4):350-91. doi: 10.6004/jnccn.2009.0027. No abstract available. PMID 19406039
- [Background] Endo I, Gonen M, Yopp AC, Dalal KM, Zhou Q, Klimstra D, D'Angelica M, DeMatteo RP, Fong Y, Schwartz L, Kemeny N, O'Reilly E, Abou-Alfa GK, Shimada H, Blumgart LH, Jarnagin WR. Intrahepatic cholangiocarcinoma: rising frequency, improved survival, and determinants of outcome after resection. Ann Surg. 2008 Jul;248(1):84-96. doi: 10.1097/SLA.0b013e318176c4d3. PMID 18580211
- [Background] Hyder O, Hatzaras I, Sotiropoulos GC, Paul A, Alexandrescu S, Marques H, Pulitano C, Barroso E, Clary BM, Aldrighetti L, Ferrone CR, Zhu AX, Bauer TW, Walters DM, Groeschl R, Gamblin TC, Marsh JW, Nguyen KT, Turley R, Popescu I, Hubert C, Meyer S, Choti MA, Gigot JF, Mentha G, Pawlik TM. Recurrence after operative management of intrahepatic cholangiocarcinoma. Surgery. 2013 Jun;153(6):811-8. doi: 10.1016/j.surg.2012.12.005. Epub 2013 Mar 15. PMID 23499016
- [Background] Tabrizian P, Jibara G, Hechtman JF, Franssen B, Labow DM, Schwartz ME, Thung SN, Sarpel U. Outcomes following resection of intrahepatic cholangiocarcinoma. HPB (Oxford). 2015 Apr;17(4):344-51. doi: 10.1111/hpb.12359. Epub 2014 Nov 14. PMID 25395176
- [Background] Wang Y, Li J, Xia Y, Gong R, Wang K, Yan Z, Wan X, Liu G, Wu D, Shi L, Lau W, Wu M, Shen F. Prognostic nomogram for intrahepatic cholangiocarcinoma after partial hepatectomy. J Clin Oncol. 2013 Mar 20;31(9):1188-95. doi: 10.1200/JCO.2012.41.5984. Epub 2013 Jan 28. PMID 23358969
- [Background] Doussot A, Gonen M, Wiggers JK, Groot-Koerkamp B, DeMatteo RP, Fuks D, Allen PJ, Farges O, Kingham TP, Regimbeau JM, D'Angelica MI, Azoulay D, Jarnagin WR. Recurrence Patterns and Disease-Free Survival after Resection of Intrahepatic Cholangiocarcinoma: Preoperative and Postoperative Prognostic Models. J Am Coll Surg. 2016 Sep;223(3):493-505.e2. doi: 10.1016/j.jamcollsurg.2016.05.019. Epub 2016 Jun 11. PMID 27296525
- [Background] Gupta R, Gupta J. Strategies to improve survival of patients with intrahepatic cholangiocarcinoma undergoing liver transplantation. Hepatology. 2017 May;65(5):1777-1778. doi: 10.1002/hep.28994. Epub 2017 Feb 3. No abstract available. PMID 27997682
- [Background] Rana A, Hong JC. Orthotopic liver transplantation in combination with neoadjuvant therapy: a new paradigm in the treatment of unresectable intrahepatic cholangiocarcinoma. Curr Opin Gastroenterol. 2012 May;28(3):258-65. doi: 10.1097/MOG.0b013e32835168db. PMID 22333563
- [Background] Sapisochin G, Facciuto M, Rubbia-Brandt L, Marti J, Mehta N, Yao FY, Vibert E, Cherqui D, Grant DR, Hernandez-Alejandro R, Dale CH, Cucchetti A, Pinna A, Hwang S, Lee SG, Agopian VG, Busuttil RW, Rizvi S, Heimbach JK, Montenovo M, Reyes J, Cesaretti M, Soubrane O, Reichman T, Seal J, Kim PT, Klintmalm G, Sposito C, Mazzaferro V, Dutkowski P, Clavien PA, Toso C, Majno P, Kneteman N, Saunders C, Bruix J; iCCA International Consortium. Liver transplantation for "very early" intrahepatic cholangiocarcinoma: International retrospective study supporting a prospective assessment. Hepatology. 2016 Oct;64(4):1178-88. doi: 10.1002/hep.28744. Epub 2016 Aug 24. PMID 27481548
- [Background] Goldstein RM, Stone M, Tillery GW, Senzer N, Levy M, Husberg BS, Gonwa T, Klintmalm G. Is liver transplantation indicated for cholangiocarcinoma? Am J Surg. 1993 Dec;166(6):768-71; discussion 771-2. doi: 10.1016/s0002-9610(05)80696-8. PMID 8273866
- [Background] Pichlmayr R, Weimann A, Oldhafer KJ, Schlitt HJ, Klempnauer J, Bornscheuer A, Chavan A, Schmoll E, Lang H, Tusch G, et al. Role of liver transplantation in the treatment of unresectable liver cancer. World J Surg. 1995 Nov-Dec;19(6):807-13. doi: 10.1007/BF00299775. PMID 8553670
- [Background] Becker NS, Rodriguez JA, Barshes NR, O'Mahony CA, Goss JA, Aloia TA. Outcomes analysis for 280 patients with cholangiocarcinoma treated with liver transplantation over an 18-year period. J Gastrointest Surg. 2008 Jan;12(1):117-22. doi: 10.1007/s11605-007-0335-4. Epub 2007 Oct 26. PMID 17963015
- [Background] Darwish Murad S, Kim WR, Harnois DM, Douglas DD, Burton J, Kulik LM, Botha JF, Mezrich JD, Chapman WC, Schwartz JJ, Hong JC, Emond JC, Jeon H, Rosen CB, Gores GJ, Heimbach JK. Efficacy of neoadjuvant chemoradiation, followed by liver transplantation, for perihilar cholangiocarcinoma at 12 US centers. Gastroenterology. 2012 Jul;143(1):88-98.e3; quiz e14. doi: 10.1053/j.gastro.2012.04.008. Epub 2012 Apr 12. PMID 22504095
- [Background] Marchan EM, Landry JC. Neoadjuvant chemoradiation followed by orthotopic liver transplantation in cholangiocarcinomas: the emory experience. J Gastrointest Oncol. 2016 Apr;7(2):248-54. doi: 10.3978/j.issn.2078-6891.2015.117. PMID 27034793
- [Background] Schule S, Altendorf-Hofmann A, Utess F, Rauchfuss F, Freesmeyer M, Knosel T, Dittmar Y, Settmacher U. Liver transplantation for hilar cholangiocarcinoma--a single-centre experience. Langenbecks Arch Surg. 2013 Jan;398(1):71-7. doi: 10.1007/s00423-012-1007-8. Epub 2012 Oct 9. PMID 23053456
- [Background] Hong JC, Petrowsky H, Kaldas FM, Farmer DG, Durazo FA, Finn RS, Saab S, Han SH, Lee P, Markovic D, Lassman C, Hiatt JR, Busuttil RW. Predictive index for tumor recurrence after liver transplantation for locally advanced intrahepatic and hilar cholangiocarcinoma. J Am Coll Surg. 2011 Apr;212(4):514-20; discussion 520-1. doi: 10.1016/j.jamcollsurg.2010.12.005. PMID 21463781
- [Background] Rea DJ, Heimbach JK, Rosen CB, Haddock MG, Alberts SR, Kremers WK, Gores GJ, Nagorney DM. Liver transplantation with neoadjuvant chemoradiation is more effective than resection for hilar cholangiocarcinoma. Ann Surg. 2005 Sep;242(3):451-8; discussion 458-61. doi: 10.1097/01.sla.0000179678.13285.fa. PMID 16135931
- [Background] Sudan D, DeRoover A, Chinnakotla S, Fox I, Shaw B Jr, McCashland T, Sorrell M, Tempero M, Langnas A. Radiochemotherapy and transplantation allow long-term survival for nonresectable hilar cholangiocarcinoma. Am J Transplant. 2002 Sep;2(8):774-9. doi: 10.1034/j.1600-6143.2002.20812.x. PMID 12243499
- [Background] Meyer CG, Penn I, James L. Liver transplantation for cholangiocarcinoma: results in 207 patients. Transplantation. 2000 Apr 27;69(8):1633-7. doi: 10.1097/00007890-200004270-00019. PMID 10836374
- [Background] Robles R, Figueras J, Turrion VS, Margarit C, Moya A, Varo E, Calleja J, Valdivieso A, Valdecasas JC, Lopez P, Gomez M, de Vicente E, Loinaz C, Santoyo J, Fleitas M, Bernardos A, Llado L, Ramirez P, Bueno FS, Jaurrieta E, Parrilla P. Spanish experience in liver transplantation for hilar and peripheral cholangiocarcinoma. Ann Surg. 2004 Feb;239(2):265-71. doi: 10.1097/01.sla.0000108702.45715.81. PMID 14745336
- [Background] Hong JC, Jones CM, Duffy JP, Petrowsky H, Farmer DG, French S, Finn R, Durazo FA, Saab S, Tong MJ, Hiatt JR, Busuttil RW. Comparative analysis of resection and liver transplantation for intrahepatic and hilar cholangiocarcinoma: a 24-year experience in a single center. Arch Surg. 2011 Jun;146(6):683-9. doi: 10.1001/archsurg.2011.116. PMID 21690444
- [Background] Jain A, Javle M. Molecular profiling of biliary tract cancer: a target rich disease. J Gastrointest Oncol. 2016 Oct;7(5):797-803. doi: 10.21037/jgo.2016.09.01. PMID 27747093
- [Background] Jain A, Kwong LN, Javle M. Genomic Profiling of Biliary Tract Cancers and Implications for Clinical Practice. Curr Treat Options Oncol. 2016 Nov;17(11):58. doi: 10.1007/s11864-016-0432-2. PMID 27658789
- [Background] Javle M, Bekaii-Saab T, Jain A, Wang Y, Kelley RK, Wang K, Kang HC, Catenacci D, Ali S, Krishnan S, Ahn D, Bocobo AG, Zuo M, Kaseb A, Miller V, Stephens PJ, Meric-Bernstam F, Shroff R, Ross J. Biliary cancer: Utility of next-generation sequencing for clinical management. Cancer. 2016 Dec 15;122(24):3838-3847. doi: 10.1002/cncr.30254. Epub 2016 Sep 13. PMID 27622582
- [Background] De Martin E, Rayar M, Golse N, Dupeux M, Gelli M, Gnemmi V, Allard MA, Cherqui D, Sa Cunha A, Adam R, Coilly A, Antonini TM, Guettier C, Samuel D, Boudjema K, Boleslawski E, Vibert E. Analysis of Liver Resection Versus Liver Transplantation on Outcome of Small Intrahepatic Cholangiocarcinoma and Combined Hepatocellular-Cholangiocarcinoma in the Setting of Cirrhosis. Liver Transpl. 2020 Jun;26(6):785-798. doi: 10.1002/lt.25737. PMID 32090444
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Lunsford KE, Javle M, Heyne K, Shroff RT, Abdel-Wahab R, Gupta N, Mobley CM, Saharia A, Victor DW, Nguyen DT, Graviss EA, Kaseb AO, McFadden RS, Aloia TA, Conrad C, Li XC, Monsour HP, Gaber AO, Vauthey JN, Ghobrial RM; Methodist-MD Anderson Joint Cholangiocarcinoma Collaborative Committee (MMAJCCC). Liver transplantation for locally advanced intrahepatic cholangiocarcinoma treated with neoadjuvant therapy: a prospective case-series. Lancet Gastroenterol Hepatol. 2018 May;3(5):337-348. doi: 10.1016/S2468-1253(18)30045-1. Epub 2018 Mar 13. PMID 29548617